CLINICAL TRIAL: NCT01936532
Title: Phase II Trial Studying the Efficacy of a Triplet Combination of MLN9708, Lenalidomide and Dexamethasone as Induction Prior to, and as Consolidation After High-dose Therapy With Peripheral Stem Cell Transplantation Followed by MLN9708 Maintenance in the Initial Management of Multiple Myeloma in Patients Younger Than 66 Years
Brief Title: Safety and Efficacy Study of a Triplet Combination of MLN9708, Lenalidomide and Dexamethasone in the Initial Management of Multiple Myeloma (IFM2013-06)
Acronym: IFM2013-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC12_0447; 2013-001443-31 (EudraCT Number)
Record Dates: First submitted 2013-07-29; First posted 2013-09-06 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Newly Diagnosed Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- assessment of treatment lenalidomide, dexamethasone,MLN9708 (Experimental)
  Interventions: Drug: MLN9708; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: MLN9708 — Induction therapy Patients will receive 3 cycles of induction therapy with MLN9708 (4 mg) on Days 1, 8 and 15, plus Lenalidomide (25 mg) on Days 1 through 21 and Dexamethasone (40 mg) on Days 1, 8, 15 and 22 of a 28-day cycle.
  Consolidation therapy
  * Early consolidation (consolidation part 1) will comprise 2 cycles of MRD identical to induction therapy.
  * Late consolidation (consolidation part 2) will consist in 6 additional cycles of MLN9708 (4 mg on Days 1, 8 and 15) plus lenalidomide (25 mg on Days 1 through 21) of a 28-day cycle.
  Maintenance therapy MLN9708 monotherapy (4 mg/day), will be given on days 1, 8 and 15 of a 28 day cycle, during 12 months.
Drug: Lenalidomide
Drug: Dexamethasone

SUMMARY:
This is a phase II, multicenter, open-label study to evaluate the safety and efficacy of MLN9708 in combination with Lenalidomide and Dexamethasone in patients with newly diagnosed multiple myeloma. The patient population will consist of adult men and women younger than 66 years, who have a confirmed diagnosis of MM who meet eligibility criteria.

Following the screening period, patients will be enrolled and treated then, they will receive induction therapy (3 cycles), a systematic Peripheral Blood Stem Cell harvest. After Peripheral Blood Stem Cell Transplantation, patient will enter in the consolidation phase (early and late one) 2 months after transplantation. Finally, patients follow a Maintenance therapy (start 1 month after the last cycle of consolidation) during 12 months.

ELIGIBILITY:
Inclusion criteria

1. Male or female patients ≥ 18 years and ≤ 65 years at the time
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
3. Patients diagnosed with multiple myeloma
4. Subjects must have symptomatic myeloma with CRAB criteria.
5. Subjects must have measurable disease requiring systemic therapy defined by serum M-component ≥ 5g/l, urine M-component ≥ 200 mg/24h or serum FLC ≥ 100 mg/l.
6. Subjects must not have been treated previously with any systemic therapy for multiple myeloma. 7.Subjects must be eligible for high dose therapy.

8.Life expectancy ≥ 3 months.9.ECOG performance status 0, 1 or 2. 10.Patients must meet the following clinical laboratory criteria

* Adequate hepatic function, with serum ALT and AST ≤ 3 times the upper limit of normal and serum direct bilirubin ≤ 1.5 times the upper limit of normal within 14 days prior to enrolment.
* Absolute neutrophil count (ANC) ≥ 1.0 × 109/L within 14 days prior to enrollment.
* Hemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior to enrollment (subjects may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines with a wash-out period of 7 days).
* Platelet count ≥ 75 × 109/L (≥ 30 × 109/L if myeloma involvement in the bone marrow is > 50%) within 14 days prior to enrollment. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
* Calculated creatinine clearance ≥ 30 mL/minute (MDRD formula should be used for calculating creatinine clearance values: http://mdrd.com/).

  11.Female of childbearing potential:must have two negative pregnancy tests : one serum pregnancy test within 10 to 14 days prior to therapy and one urine pregnancy test within 24 hours before starting study drug.

must agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 3 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.

12.Male patients, even if surgically sterilized, must agree to not father a child and agree to use a latex condom during therapy and for 3 months after the last dose of study drug, even if they have had a successful vasectomy, if their partner is of childbearing potential.

13.Affiliation number to National Health Care System.

Exclusion Criteria:

1. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test within 24 hours before first dose of study drug.
2. Evidence of mucosal or internal bleeding and/or platelet refractory.
3. Prior myeloma systemic therapy.
4. Major surgery within 14 days before first dose of study drug.
5. Radiotherapy within 14 days before first dose of study drug. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708.
6. Treatment by corticosteroids if exceed the equivalent of 160 mg of dexamethasone within 14 days before first dose of study drug.
7. Subjects not eligible for high dose therapy.
8. Growth factors within 7 days prior to enrolment.
9. Transfusion within 3 days prior to enrolment.
10. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to first dose of study drug.
11. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before first dose of study drug.
12. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within 6 months.
13. Systemic treatment, within 14 days before first dose of study drug, with strong inhibitors of CYP1A2, strong inhibitors of CYP3A or strong CYP3A inducers, or use of Ginkgo biloba or St. John's wort.
14. Ongoing or active systemic infection, known human immunodeficiency virus positive, known active hepatitis B virus hepatitis, or known active hepatitis C virus hepatitis.
15. Co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
16. Psychiatric illness/social situation that would limit compliance with study requirements.
17. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
18. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
19. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or GI procedure that could interfere with the oral absorption or tolerance of treatment.
20. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
21. Patient has significant neuropathy within 14 days prior to enrolment.
22. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrolment.
23. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.
24. Participation in clinical trials with other investigational agents not included in this trial, within 21days of the start of this trial and throughout the duration of this trial.
25. Failure to have fully recovered from the reversible effects of prior chemotherapy.
26. Central nervous system involvement

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the stringent Complete Response (sCR) rate of the combination of MLN9708, Lenalidomide and Dexamethasone in newly diagnosed multiple myeloma (MM) patients after extended consolidation therapy | sixteen months

SECONDARY OUTCOMES:
To evaluate the overall response rate after induction therapy | after 63 days
To evaluate the safety Evaluate the safety | after 63 days
  Descriptive statistics of treatment duration cumulative dose, dose intensity and relative dose intensity will be presented.
  Treatment emergent adverse events will be summarized by period (induction, consolidation and maintenance) and overall.
  Overall adverse events will be summarized by system organ class and preferred term and by severity (worst toxicity grade owing to the NCI CTCAE v4.0).
To evaluate the quality of stem cell harvest | after 84 days
  according to institutional practice, participants must collect a minimum CD34 count of > 5x106 cells/kg. In case of insufficient collection, collection of a minimum CD34 count of > 2x106 cells/kg will be allowed.
  Thus the number of cells collected will be evaluated
To evaluate the overall response rate after high-dose therapy (prior to consolidation) | after 84 days
To evaluate the overall response rate after consolidation therapy | after 270 days
To evaluate the feasibility of maintenance with MLN9708 | after 270 days
  number of dose
To evaluate duration of response, progression-free and overall survival | five years and a half

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MOREAU, Principal Investigator — Nantes University Hospital
Locations (10):
- France (10):
  - CHRU - Hôpital du Haut Lévêque, Bordeaux
  - CHRU Dijon, Dijon
  - Centre hospitalier départemental Vendée, La Roche-sur-Yon
  - CHRU - Hôpital Claude Huriez, Lille
  - Nantes University Hospital, Nantes
  - Hôpital Saint-Antoine, Paris
  - Centre Hospitalier Lyon sud, Pierre-Bénite
  - Pole IUC Oncopole CHU, Toulouse
  - CHRU - Hôpital Bretonneau, Tours
  - CHRU - Hôpitaux de Brabois, Vandœuvre-lès-Nancy